CLINICAL TRIAL: NCT01107847
Title: Measurement of Regional Lung Opening and Closing Pressures in Patients With Acute Lung Injury Using Electrical Impedance Tomography
Brief Title: Regional Lung Opening and Closing Pressures in Patients With Acute Lung Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Prof. Dr. Jens Scholz, University of Schleswig-Holstein
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UKSH ROP/RCP
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-03

CONDITIONS: Acute Lung Injury
Keywords: electrical impedance tomography; EIT; acute lung injury; regional lung opening pressure; regional lung closing pressure
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: low flow pressure volume manoeuvre — In all patients a standard low flow pressure volume manoeuvre is applied by a respirator with a constant gas flow of 4 l/min starting at a zero end-expiratory pressure up to a tidal volume of 2 l or until a maximum airway pressure of 35 cm H2O was reached.

SUMMARY:
The purpose of this study is the measurement of regional opening and closing pressures of lung tissue by electrical impedance tomography in lung healthy and patients with acute lung injury. These values might help the setting of positive endexpiratory pressure during artificial ventilation to avoid the cyclic opening and closing of alveoli.

DETAILED DESCRIPTION:
During artificial ventilation the cyclic opening and closing of alveoli during artificial ventilation results in patients with acute lung injury (ALI) in a higher mortality. A positive endexpiratory pressure (PEEP) is applied with the intention to avoid these cyclic opening and closing of alveoli. The distribution of ventilation in patients with ALI is extremely inhomogeneous, consequently there are different regional opening pressures needed to open up the alveoli and avoid closing. Finding the best level of PEEP in patients with injured lungs to avoid atelectasis and alveolar strain induced by inadequately high or low PEEP levels is a challenge.

The purpose of this study is to develop a protocol for measuring regional opening and closing pressures using the method of electrical impedance tomography in lung healthy and ALI patients. A ventilator setting guided by regional opening and closing pressures might help reducing the impairment of the lung by artificial ventilation.

ELIGIBILITY:
Inclusion Criteria:

* artificial ventilation
* acute lung injury / healthy lung (control group)

Exclusion Criteria:

* pregnancy
* Cerebral trauma / surgery
* Age < 18 years
* instable cardiovascular disease
* instable chest wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)

PRIMARY OUTCOMES:
Measurement of regional lung opening pressures | one year
  For the measurement of regional opening pressures in lung healthy and acute lung injury an inspiratory low flow manoeuvre with synchronous measurement of regional ventilation and airway pressure is performed. The regional opening pressures are defined as the airway pressure to the point were the regional lung areas open up.

SECONDARY OUTCOMES:
Measurement of regional closing pressures | one year
  For the measurement of regional closing pressures in lung healthy and acute lung injury an expiratory low flow manoeuvre with synchronous measurement of regional ventilation and airway pressure is performed. The regional closing pressures are defined as the airway pressure to the point were the regional lung areas start closing.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Scholz, M.D., Study Chair — University Medical Center of Schleswig-Holstein, Campus Kiel, Department of Anesthesiology and Intensive Care Medicine
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, University Medical Center of Schleswig-Holstein, Campus Kiel, Kiel, Germany

REFERENCES:
- [Background] Caironi P, Cressoni M, Chiumello D, Ranieri M, Quintel M, Russo SG, Cornejo R, Bugedo G, Carlesso E, Russo R, Caspani L, Gattinoni L. Lung opening and closing during ventilation of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2010 Mar 15;181(6):578-86. doi: 10.1164/rccm.200905-0787OC. Epub 2009 Nov 12. PMID 19910610
- [Background] Wrigge H, Zinserling J, Muders T, Varelmann D, Gunther U, von der Groeben C, Magnusson A, Hedenstierna G, Putensen C. Electrical impedance tomography compared with thoracic computed tomography during a slow inflation maneuver in experimental models of lung injury. Crit Care Med. 2008 Mar;36(3):903-9. doi: 10.1097/CCM.0B013E3181652EDD. PMID 18431279
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669